CLINICAL TRIAL: NCT03938051
Title: Effects of Multicomponent Exercise on Mild Cognitive Impairment In Elderly Population ,a Randomized Control Trial
Brief Title: Multi-component Exercise on Mild Cognitive Impairment In Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Hafsah Gul Khattak
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Exercise; Mild Cognitive Impairment; Elderly Population
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Multi-component intervention
  Interventions: Other: Experimental group
- Control group (Experimental): treadmill walk
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — Multicomponent intervention for twice weekly 55-60 minutes 6 weeks
  Arms: Experimental group
Other: Control group — 20 minutes treadmill walk thrice weekly, 5-7 /10 subjective rate of perceived exertion
  Arms: Control group

SUMMARY:
Participants will be randomized to exercise intervention and control groups, for 6 weeks. The participants will be examined for following test Mini mental state examination, Trail making test A and B, MOCA. The intervention will consist of twice weekly, 55- 60 minute exercise session for experimental group The participants of control group will receive 20 minutes treadmill walk thrice weekly. Participants will walk at constant pace with zero inclination such that a subjective rate of perceived of 5 to 7 points on the ten-point Borg scale will be reached. Assessment of both groups will be done on first session and on last session.

DETAILED DESCRIPTION:
Elderly, old person and senior citizen are all the terms generally used for geriatric population. According to WHO, most developed countries have accepted the chronological age of 65 years as definition of elderly or older population which cannot be applied to developing third world countries as the life expectancy is between 60 to 70 years. The United Nation agreed cutoff is 60+ years to refer to old age. Adding to difficulty of defining actual birth dates is often unknown in some areas because many people do not have official birth records.

Aging is characterized by gradual irreversible changes in structure and function of an individual that occur as a result of the passage of time. It is additionally subject to the developments by which general public understands maturity. It is associated with declines in different systems of body, resulting in an impaired capacity to perform daily activities placing a large economic burden on society. Life of the elderly is characterized by a high risk of multimorbidity accompanied by a high prevalence of cognitive impairment short of dementia. A decline in cognitive abilities, such as perception, reasoning, and memory, is part of the normal cognitive aging process. It is a process that is genetically defined and environmentally modulated. In fact, advancing age is the major risk factor for a number of chronic diseases in humans. A decrease in cognitive performance in older adults is predominant in most individuals. During next 40 years, it is anticipated that there will be an epidemic of dementia worldwide, with a 3- to 4-fold increase in the number of prevalent cases owing to longer life expectancies and demographic changes. Attention is turning toward identification of preclinical disease and development of treatments to prevent or delay the onset of dementia. Cognitive impairment is a health problem that almost concerns to every second elderly person.

There is of evidence from epidemiological studies, experimental trials, and basic neurosciences that suggesting that cognitive decline related to aging can be cut off by different intellectual activities which makes you less prone to cognitive problems faced at later ages. There is always a debate whether cognitive mental activities are more better or physical activity is better solution for these age related cognitive decline .Some studies showed that cognitive training is effective when cognitive skills are practiced.

Cognitive decline due to aging leads to functional limitation and disability which leaves the society with a huge economic burden. That is why, intervention and plan should be designed to lessen this economic burden furthermore maintain and control epidemics like dementia and other cognitive disorders. Physical activity has shown tremendous results in improving cognition function in healthy older adults and as well as in older adults affected with cognitive diseases and disorders. Evidence from epidemiological studies shows that physical activity of high levels and for longer follow-ups showed better results in decreasing the likelihood of developing cognitive impairments as compared to people with low levels of physical activity .Therefore, it is hypothesized that physical activity plays an important role in alleviating cognitive decline in older adults. Physical movement has been appeared to have an intense up regulating impact on neurogenesis and to result in increased concentration of brain derived neurotropic factor.

Despite of the beneficial effects observed in cognitive outcomes with aerobic exercise training in Previous studies aerobic exercise was associated with progress in neurocognitive functions in older adults whether cognitive impairment is present or not . A study conducted in 2012 reported significant improvements in memory domain and few other studies showed significant improvements in executive function after following aerobic training protocol. But there was lack of consistent evidence to show the beneficial effects of aerobic training on cognition in elderly population. Many other researchers focused on resistive training exercises for improving cognitive and memory functions.With advancement of time and technology newer exercise techniques and modalities have been developed to maximize functional capacities of older adults. In these days of development multi-component exercises is a new combination of training exercise in which aerobic, resistance training is combined with balance ,coordination, flexibility to decrease disability in older adults.Multi-component is the most effective approach in addressing functional capacity in frail older adults and limiting disability.Functional benefits of this exercise are well established ,however evidence is less consistent regarding cognitive gains associated with multi-component exercise training. A study reported that aerobic and resistance training combined has better gains in working memory as compared to aerobic training alone.

In the light of literature review studies were conducted to determine the effects of different types of physical activity on cognition of elderly people and in prevention of decreasing cognitive levels in elderly people. The impact of exercises including aerobic training, resistive training, aerobic training versus stretching, resistive training versus stretching, resistive training with no intervention were previously examined however, results were less clear and consistent.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women
* Mini-Mental State Examination (MMSE) score 18- 23 (mild cognitive impairment)

Exclusion Criteria:

* Had current medical condition for which exercise is contraindicated
* Had neurodegenerative disease /stroke
* Oncologic patient with active treatment with chemotherapy
* Patient with arterial diseases in the past 12 months

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Mini mental state examination (MMSE) | 6 week
  Changes from the Baseline, Mini mental state examination (MMSE): used to screen for cognitive impairment in elderly. It is as 30-point questionnaire. The reliability of the MMSE, ranging from 0.76 to 0.90.
Trail making test (TMT) A & B | 6 week
  Changes from the Baseline, Trail making test (TMT) A & B: It is a test of visual attention and task switching. It provides information about visual search speed, speed of processing and executive function. The test reliability for TMT (A -B) is 0.82 and 0.93. Time will be measured in seconds
Montreal cognitive assessment (MoCA) | 6 week
  Changes from the Baseline, Montreal cognitive assessment (MoCA): it is used widely for screening cognitive impairment.The test re-test reliability for MOCA is 0.966. Scoring. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal. In a study, normal people scored an average of 27.4; people with mild cognitive impairment (MCI) scored an average of 22.1; people with Alzheimer's disease scored an average of 16.2.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No